CLINICAL TRIAL: NCT04330612
Title: Perioperative Family Updates Reduce Anxiety and Improve Satisfaction: A Randomized Controlled Trial
Brief Title: Perioperative Family Updates Reduce Anxiety and Improve Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont Medical Center (Other)
Responsible Party: Principal Investigator, Lindsay Howe, Primary Researcher, University of Vermont Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CHRMS 16-642
Record Dates: First submitted 2020-03-29; First posted 2020-04-01 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Family Members; Anxiety; Satisfaction
MeSH Terms: conditions — Anxiety Disorders; Personal Satisfaction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): In the control pathway, the surgeons communicated with the family only once near the completion of the procedure.
- Intervention (Experimental): In the intervention group, the families received additional standardized electronic updates via pagers.
  Interventions: Other: Perioperative Updates

INTERVENTIONS:
Other: Perioperative Updates — In the intervention group, the families received additional standardized electronic updates via pagers at three pivotal moments: 1) Initial skin incision has been made; 2) Critical part of the case is completed and closure has begun; and, 3) Closure is complete, and patient will be transferred to the recovery room when ready.
  Arms: Intervention

SUMMARY:
This study was a randomized control trial conducted to determine if frequent, standardized updates affect anxiety and satisfaction of family members. Additionally, the investigators aimed to determine if the length of the surgical procedure effects the satisfaction with updates.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing inpatient arthroplasty, orthopaedic spine, or orthopaedic trauma procedures

Exclusion Criteria:

* Age under 18
* Non-English speaking patients or families
* Patients with families that would not be waiting in the hospital during the perioperative period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Likert Score (0-5) of level of overall satisfaction | Overall satisfaction levels measured throughout the perioperative period (up to 8.4 hours), reported at the time of final surgeon-family update. This update occurred at or near the end of the surgical procedure.
  Likert Score (0-5) of level of overall satisfaction of family members throughout the perioperative period
Likert Score (0-5) of anxiety level | Anxiety levels measured throughout the perioperative period (up to 8.4 hours), reported at the time of final surgeon-family update. This update occurred at or near the end of the surgical procedure.
  Likert Score (0-5) of anxiety level of family members throughout the perioperative period
Likert Score (0-5) of level of satisfaction with perioperative updates | Satisfaction with perioperative updates measured throughout the perioperative period (up to 8.4 hours), reported at the time of final surgeon-family update. This update occurred at or near the end of the surgical procedure.
  Likert Score (0-5) of level of satisfaction of family members with perioperative updates throughout the perioperative period

SECONDARY OUTCOMES:
Spearman correlation between length of procedure and Likert score of anxiety level | Procedure time defined as the time the patient enters the operating room to the time the patient exits the operating room. Anxiety levels measured throughout the perioperative period (up to 8.4 hours), reported at the time of final surgeon update.
  Spearman correlation between length of procedure and Likert score (0-5) of anxiety level of family members throughout the perioperative period
Spearman correlation between length of procedure and Likert score of overall satisfaction | Procedure time defined as the time the patient enters the operating room to the time the patient exits the operating room. Satisfaction level measured throughout the perioperative period (up to 8.4 hours), reported at the time of final surgeon update.
  Spearman correlation between length of procedure and Likert score (0-5) of overall satisfaction level of family members throughout the perioperative period
Spearman correlation between length of procedure and Likert score of satisfaction with perioperative updates | Procedure time defined as the time the patient enters the operating room to the time the patient exits the operating room. Satisfaction level measured throughout the perioperative period (up to 8.4 hours), reported at the time of final surgeon update.
  Spearman correlation between length of procedure and Likert score of family member satisfaction with perioperative updates

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-20): https://cdn.clinicaltrials.gov/large-docs/12/NCT04330612/Prot_SAP_000.pdf